CLINICAL TRIAL: NCT03439657
Title: Immunogenicity and Safety Study of GSK Biologicals' Herpes Zoster Vaccine GSK1437173A When Co-administered With Prevenar13 in Adults Aged 50 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 204487; 2017-001220-22 (EudraCT Number)
Record Dates: First submitted 2018-02-12; First posted 2018-02-20 (Actual); Results first posted 2021-03-18 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-10

CONDITIONS: Herpes Zoster
Keywords: HZ; Safety; Immunogenicity; Shingles; Adults; Prevenar 13
MeSH Terms: conditions — Herpes Zoster | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Co-Ad Group (Experimental): Adults aged ≥50 years of age who received the first dose of GSK1437173A and one dose of Prevenar13 at Day 1 and the second dose of GSK1437173A at Month 2. Both vaccines were administered intramuscularly, GSK1437173A was administered in the deltoid muscle of the non-dominant arm, while Prevenar13 was administered in the deltoid muscle of the dominant arm
  Interventions: Biological: HZ/su vaccine GSK1437173A; Biological: Prevenar13
- Control Group (Active Comparator): Adults aged ≥50 years of age who received one dose of Prevenar13 at Day 1, the first dose of GSK1437173A at Month 2 and the second dose of GSK1437173A at Month 4. Both vaccines were administered intramuscularly, GSK1437173A was administered in the deltoid muscle of the non-dominant arm, while Prevenar13 was administered in the deltoid muscle of the dominant arm
  Interventions: Biological: HZ/su vaccine GSK1437173A; Biological: Prevenar13

INTERVENTIONS:
Biological: HZ/su vaccine GSK1437173A — 2 doses of 0.5 mL of the vaccine in a 0,2 Months schedule. Administered by intramuscular injection into the deltoid muscle of the non-dominant arm.
Biological: Prevenar13 — 1 dose of 0.5 mL of the vaccine. Administered by intramuscular injection into the deltoid muscle of the dominant arm.
  Other Names: PCV13

SUMMARY:
The purpose of this study is to assess immunogenicity and safety of GSK Biologicals' HZ vaccine when its first dose is co-administered with a pneumococcal polysaccharide conjugate vaccine (Prevenar13) in adults aged ≥50 YOA, as compared to the control group where the two HZ/su doses are administered subsequent to Prevenar13.

DETAILED DESCRIPTION:
Following the initial approval of the GlaxoSmithKline (GSK) Biologicals' HZ/su vaccine, the protocol was amended to indicate that the trademark is Shingrix. In addition, the term "candidate" vaccine has been replaced by "study" vaccine throughout the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performance of any study specific procedure.
* A male or female, aged ≥50 YOA at the time of the first vaccination with the study vaccine(s).
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines during the period starting 30 days before the first dose of study vaccines (Day -30 to Day 1), or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular (IM) injection unsafe.
* Use or anticipated use of immunosuppressants or other immune-modifying drugs during the period starting six months prior to study start and during the whole study period. This includes chronic administration of corticosteroids (>14 consecutive days of prednisone at a dose of ≥20 mg/day [or equivalent]), long-acting immune modifying agents or immunosuppressive/cytotoxic therapy. Inhaled, topical and intra-articular corticosteroids are allowed.
* Administration or planned administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of study vaccine administration. This includes any type of vaccine such as (but not limited to) live, inactivated and subunit vaccines.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Previous and/or planned administration of an HZ or VZV vaccine other than the study vaccine during the study period.
* History of HZ.
* History of documented pneumococcal infection within 5 previous years.
* Prior receipt of any pneumococcal vaccine or planned use during the study period, other than the study vaccines.
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Acute disease and/or fever at the time of enrollment.

  * Fever is defined as temperature ≥ 38.0°C/100.4°F. The preferred location for measuring temperature in this study will be the oral cavity.
  * Subjects with a minor illness without fever may, be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions before 2 months after the last dose of study vaccine.
* Any person with cerebrospinal fluid (CSF) leaks, cochlear implants, chronic renal failure, nephrotic syndrome and functional or anatomic asplenia.
* Any medical condition that in the judgment of the investigator would prevent the subject from participating in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 913 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (3):
  - GSK Investigational Site, Marlborough, Massachusetts
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
- Canada (2):
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Sherbrooke, Quebec
- Estonia (3):
  - GSK Investigational Site, Rakvere
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (5):
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate

REFERENCES:
- [Derived] Min JY, Mwakingwe-Omari A, Riley M, Molo LY, Soni J, Girard G, Danier J. The adjuvanted recombinant zoster vaccine co-administered with the 13-valent pneumococcal conjugate vaccine in adults aged >/=50 years: A randomized trial. J Infect. 2022 Apr;84(4):490-498. doi: 10.1016/j.jinf.2021.12.033. Epub 2021 Dec 25. PMID 34963639

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 4 countries (Canada, Estonia, Germany & United States)
Pre-assignment Details: Out of 913 subjects enrolled in the study, 1 subject violated protocol prior to randomization. 912 subjects were vaccinated and included in the Exposed Set, 901 subjects completed the study.
Period: Overall Study
Arm/Group | Co-Ad Group | Control Group
Started | 449 | 463
Completed | 442 | 459
Not Completed | 7 | 4
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Consent withdrawal, not due to an Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Co-Ad Group | Control Group | Total
Number analyzed (Participants) | 449 | 463 | 912
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.1 (8.3) | 63.2 (8.4) | 63.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 284 | 543
  Male | 190 | 179 | 369
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 1 | 0 | 1
  Black Or African American | 8 | 8 | 16
  Mixed Origin | 0 | 2 | 2
  White - Arabic / North African Heritage | 1 | 1 | 2
  White - Caucasian / European Heritage | 439 | 452 | 891

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a Vaccine Response for Anti-glycoprotein E (Anti-gE) in Co-Ad Group
Description: Vaccine response rate (VRR) for Varicella Zoster Virus (VZV) anti-glycoprotein E (gE) humoral immunogenicity was determined by Enzyme Limked Immunosorbent Assay (ELISA). The VRR for anti-gE is defined as the percentage of subjects who had at least: a 4-fold increase in the anti-gE antibodies concentration as compared to the pre-vaccination anti-gE antibodies concentration, for subjects who are seropositive at baseline, or, a 4-fold increase in the anti-gE antibodies concentration as compared to the anti-gE antibodies cut-off value for seropositivity, for subjects who are seronegative at baseline.
Time Frame: One month post-dose 2 (Month 3)
Population: Analysis was performed on the Per-Protocol Set (PPS) for immunogenicity that included all evaluable subjects who met all eligibility criteria, who complied with the procedures and intervals allowed for the analysis and for whom data concerning immunogenicity outcome measures were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Co-Ad Group
Number analyzed (Participants) | 426
Percentage of subjects | 99.1 [97.6 to 99.7]

2. Primary Outcome: Anti-gE Antibody Concentrations
Description: Anti-gE antibody concentrations in terms of Geometric Mean concentrations (GMC) were determined by ELISA and expressed as milli-international units per milliliter (mIU/mL)
Time Frame: One month post-dose 2 (at Month 3 for the Co-Ad and Month 5 for the Control group).
Population: Analysis was performed on the PPS for immunogenicity that included all evaluable subjects who met all eligibility criteria, who complied with the procedures and intervals allowed for the analysis and for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: mlU/mL
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 426 | 436
mlU/mL | 54789.9 [51586.3 to 58192.4] | 59126.7 [55973.8 to 62457.1]

3. Primary Outcome: Anti-pneumococcal Antibody Titers
Description: Anti-pneumococcal antibody titers for the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F) were determined by Multiplex Opsonophagocytosis Assay (MOPA)
Time Frame: At one month post-dose 1 (Month 1)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 425 | 434
Titers
  MOPA-1 | 144.2 [120.5 to 172.6] | 151.5 [126.0 to 182.1]
  MOPA-3 | 99.8 [87.2 to 114.1] | 100.2 [88.0 to 114.1]
  MOPA-4 | 1127.2 [975.5 to 1302.5] | 1392.4 [1206.5 to 1607.0]
  MOPA-5: number analyzed (Participants) | 424 | 434
  MOPA-5 | 279.4 [231.2 to 337.7] | 292.8 [243.5 to 352.1]
  MOPA-6A | 1839.3 [1570.0 to 2154.9] | 2354.9 [2015.0 to 2752.2]
  MOPA-6B: number analyzed (Participants) | 425 | 433
  MOPA-6B | 1499.4 [1241.2 to 1811.4] | 2025.9 [1715.5 to 2392.4]
  MOPA-7F | 1981 [1735.2 to 2261.5] | 2387.5 [2112.7 to 2698.0]
  MOPA-9V | 2541.9 [2219.2 to 2911.7] | 3049.3 [2693.7 to 3451.9]
  MOPA-14: number analyzed (Participants) | 424 | 432
  MOPA-14 | 1752.6 [1505.2 to 2040.6] | 2096 [1796.6 to 2445.2]
  MOPA-18C | 1450.3 [1262.5 to 1666.1] | 1606.6 [1402.6 to 1840.4]
  MOPA-19A | 1684.9 [1477.2 to 1921.9] | 1664.3 [1465.7 to 1889.7]
  MOPA-19F | 712 [617.1 to 821.6] | 802.4 [696.2 to 924.8]
  MOPA-23F | 758.1 [644.9 to 891.2] | 925.5 [782.5 to 1094.7]

4. Primary Outcome: Adjusted Geometric Mean Concentrations (GMCs) for Anti-gE Antibody
Description: Anti-gE antibody concentrations (GMCs) adjusted for age and baseline concentrations were determined using Analysis Of Covariance (ANCOVA) model. Adjusted GMCs were expressed in milli-international units per milliliter (mIU/mL)
Time Frame: One month post-dose 2 (at Month 3 for the Co-Ad and Month 5 for the Control group).
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mlU/mL
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 435 | 426
mlU/mL | 58526.8 [55248.5 to 61999.7] | 54634.9 [51546.0 to 57909.0]
Statistical Analysis 1: Comparison: Control Group vs Co-Ad Group; Anti-gE GMCs (non-inferiority): Non-inferiority comparison between Control Group and Co-Ad Group in terms of geometric mean concentrations (GMCs) for anti-gE antibodies, one month after the administration of last vaccine dose; Test type: Non-Inferiority — Upper limit (UL) of the 95% confidence interval (CI) for the anti-gE antibodies Geometric Mean Concentration (GMC) ratio between the Control group and the Co-Ad group should be <1.5; ANCOVA; The 95% CI of the group GMCs ratio was computed using an Analysis Of Covariance (ANCOVA) model on the log10 transformation of the concentrations; GMC ratio = 1.07, 95% CI 2-sided [0.99 to 1.16]

5. Primary Outcome: Adjusted Geometric Mean Titers (GMTs) of Anti-pneumococcal Antibodies
Description: Geometric mean antibody (anti-pneumococcal antibodies: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F) titers adjusted for age and baseline concentration were determined using ANCOVA model.
Time Frame: At one month post-dose 1 (Month 1)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 433 | 425
Titers
  MOPA-1 | 147.1 [123.9 to 174.7] | 141.2 [118.7 to 167.9]
  MOPA-3: number analyzed (Participants) | 431 | 425
  MOPA-3 | 99.6 [88.1 to 112.6] | 97.3 [86.0 to 110.0]
  MOPA-4: number analyzed (Participants) | 432 | 423
  MOPA-4 | 1331.6 [1155.2 to 1535.0] | 1066.9 [924.2 to 1231.5]
  MOPA-5: number analyzed (Participants) | 433 | 423
  MOPA-5 | 278.9 [234.4 to 331.8] | 269.1 [225.8 to 320.8]
  MOPA-6A: number analyzed (Participants) | 433 | 424
  MOPA-6A | 2253.8 [1935.6 to 2624.3] | 1784.4 [1530.2 to 2080.8]
  MOPA-6B: number analyzed (Participants) | 431 | 424
  MOPA-6B | 1967.3 [1661.5 to 2329.3] | 1445.4 [1219.3 to 1713.4]
  MOPA-7F: number analyzed (Participants) | 432 | 423
  MOPA-7F | 2337.3 [2061.2 to 2650.5] | 1935.1 [1704.3 to 2197.1]
  MOPA-9V: number analyzed (Participants) | 431 | 420
  MOPA-9V | 2955.8 [2601.9 to 3357.9] | 2553.5 [2244.2 to 2905.4]
  MOPA-14: number analyzed (Participants) | 430 | 423
  MOPA-14 | 1992.3 [1718.5 to 2309.7] | 1730.7 [1491.3 to 2008.5]
  MOPA-18C: number analyzed (Participants) | 433 | 423
  MOPA-18C | 1558.9 [1363.9 to 1781.9] | 1403.8 [1226.4 to 1606.8]
  MOPA-19A: number analyzed (Participants) | 431 | 425
  MOPA-19A | 1663.5 [1474.0 to 1877.2] | 1619.2 [1433.7 to 1828.7]
  MOPA-19F: number analyzed (Participants) | 433 | 424
  MOPA-19F | 760.2 [664.8 to 869.2] | 696.4 [608.2 to 797.3]
  MOPA-23F: number analyzed (Participants) | 432 | 425
  MOPA-23F | 896.6 [765.0 to 1050.9] | 748.2 [637.6 to 878.0]
Statistical Analysis 1: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody titers (non-inferiority): Non-inferiority comparison between Control Group and Co-Ad Group in terms of geometric mean titers (GMTs) for anti-pneumococcal antibody (MOPA-1), one month after the administration of Prevnar 13 vaccine dose; Test type: Non-Inferiority — Upper limit (UL) of 95% CI for each individual pneumococcal conjugate serotype Geometric Mean Titer (GMT) ratio of the Control group over the Co-Ad group should be <2; ANCOVA; The 95% CI of the group MOPA GMT ratios was computed using an Analysis Of Covariance (ANCOVA) model on the log10 transformation of the concentrations; GMT ratio = 1.04, 95% CI 2-sided [0.82 to 1.33]
Statistical Analysis 2: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody titers (non-inferiority): Non-inferiority comparison between Control Group and Co-Ad Group in terms of geometric mean titers (GMTs) for anti-pneumococcal antibody (MOPA-3), one month after the administration of Prevnar 13 vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; ANCOVA; [statistical method as in outcome 5, analysis 1]; GMT ratio = 1.02, 95% CI 2-sided [0.86 to 1.22]
Statistical Analysis 3: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody titers (non-inferiority): Non-inferiority comparison between Control Group and Co-Ad Group in terms of geometric mean titers (GMTs) for anti-pneumococcal antibody (MOPA-4), one month after the administration of Prevnar 13 vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; ANCOVA; [statistical method as in outcome 5, analysis 1]; GMT ratio = 1.25, 95% CI 2-sided [1.02 to 1.52]
Statistical Analysis 4: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody titers (non-inferiority): Non-inferiority comparison between Control Group and Co-Ad Group in terms of geometric mean titers (GMTs) for anti-pneumococcal antibody (MOPA-5), one month after the administration of Prevnar 13 vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; ANCOVA; [statistical method as in outcome 5, analysis 1]; GMT ratio = 1.04, 95% CI 2-sided [0.81 to 1.32]
Statistical Analysis 5: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody titers (non-inferiority): Non-inferiority comparison between Control Group and Co-Ad Group in terms of geometric mean titers (GMTs) for anti-pneumococcal antibody (MOPA-6A), one month after the administration of Prevnar 13 vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; ANCOVA; [statistical method as in outcome 5, analysis 1]; GMT ratio = 1.26, 95% CI 2-sided [1.02 to 1.56]
Statistical Analysis 6: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody titers (non-inferiority): Non-inferiority comparison between Control Group and Co-Ad Group in terms of geometric mean titers (GMTs) for anti-pneumococcal antibody (MOPA-6B), one month after the administration of Prevnar 13 vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; ANCOVA; [statistical method as in outcome 5, analysis 1]; GMT ratio = 1.36, 95% CI 2-sided [1.07 to 1.73]
Statistical Analysis 7: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody titers (non-inferiority): Non-inferiority comparison between Control Group and Co-Ad Group in terms of geometric mean titers (GMTs) for anti-pneumococcal antibody (MOPA-7F), one month after the administration of Prevnar 13 vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; ANCOVA; [statistical method as in outcome 5, analysis 1]; GMT ratio = 1.21, 95% CI 2-sided [1.01 to 1.44]
Statistical Analysis 8: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody titers (non-inferiority): Non-inferiority comparison between Control Group and Co-Ad Group in terms of geometric mean titers (GMTs) for anti-pneumococcal antibody (MOPA-9V), one month after the administration of Prevnar 13 vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; ANCOVA; [statistical method as in outcome 5, analysis 1]; GMT ratio = 1.16, 95% CI 2-sided [0.97 to 1.39]
Statistical Analysis 9: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody titers (non-inferiority): Non-inferiority comparison between Control Group and Co-Ad Group in terms of geometric mean titers (GMTs) for anti-pneumococcal antibody (MOPA-14), one month after the administration of Prevnar 13 vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; ANCOVA; [statistical method as in outcome 5, analysis 1]; GMT ratio = 1.15, 95% CI 2-sided [0.94 to 1.42]
Statistical Analysis 10: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody titers (non-inferiority): Non-inferiority comparison between Control Group and Co-Ad Group in terms of geometric mean titers (GMTs) for anti-pneumococcal antibody (MOPA-18C), one month after the administration of Prevnar 13 vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; ANCOVA; [statistical method as in outcome 5, analysis 1]; GMT ratio = 1.11, 95% CI 2-sided [0.92 to 1.34]
Statistical Analysis 11: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody titers (non-inferiority): Non-inferiority comparison between Control Group and Co-Ad Group in terms of geometric mean titers (GMTs) for anti-pneumococcal antibody (MOPA-19A), one month after the administration of Prevnar 13 vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; ANCOVA; [statistical method as in outcome 5, analysis 1]; GMT ratio = 1.03, 95% CI 2-sided [0.87 to 1.22]
Statistical Analysis 12: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody titers (non-inferiority): Non-inferiority comparison between Control Group and Co-Ad Group in terms of geometric mean titers (GMTs) for anti-pneumococcal antibody (MOPA-19F), one month after the administration of Prevnar 13 vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; ANCOVA; [statistical method as in outcome 5, analysis 1]; GMT ratio = 1.09, 95% CI 2-sided [0.90 to 1.32]
Statistical Analysis 13: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody titers (non-inferiority): Non-inferiority comparison between Control Group and Co-Ad Group in terms of geometric mean titers (GMTs) for anti-pneumococcal antibody (MOPA-23F), one month after the administration of Prevnar 13 vaccine dose; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; ANCOVA; [statistical method as in outcome 5, analysis 1]; GMT ratio = 1.20, 95% CI 2-sided [0.96 to 1.50]

6. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms by Vaccine and Dose
Description: Assessed solicited local symptoms were pain, erythema and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 erythema/swelling = erythema/swelling that had spread beyond 100 millimeters (mm) of injection site. The Co-Ad Group received only 2 vaccine doses.
Time Frame: Within 7 days (Day 1 - 7) after each vaccination
Population: Analysis was performed on Exposed Set (ES) which included all subjects with at least one vaccine administration documented and who provided solicited safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 447 | 463
Participants
  Any Erythema, GSK1437173A, Dose1: number analyzed (Participants) | 447 | 0
  Any Erythema, GSK1437173A, Dose1 | 120 | 0
  Grade3 Erythema, GSK1437173A, Dose1: number analyzed (Participants) | 447 | 0
  Grade3 Erythema, GSK1437173A, Dose1 | 5 | 0
  Any Erythema, Prevenar13, Dose1 | 48 | 31
  Grade3 Erythema, Prevenar13, Dose1 | 2 | 1
  Any Pain, GSK1437173A, Dose1: number analyzed (Participants) | 447 | 0
  Any Pain, GSK1437173A, Dose1 | 332 | 0
  Grade3 Pain, GSK1437173A, Dose1: number analyzed (Participants) | 447 | 0
  Grade3 Pain, GSK1437173A, Dose1 | 25 | 0
  Any Pain, Prevenar13, Dose1 | 233 | 241
  Grade3 Pain, Prevenar13, Dose1 | 11 | 9
  Any Swelling, GSK1437173A, Dose1: number analyzed (Participants) | 447 | 0
  Any Swelling, GSK1437173A, Dose1 | 69 | 0
  Grade3 Swelling, GSK1437173A, Dose1: number analyzed (Participants) | 447 | 0
  Grade3 Swelling, GSK1437173A, Dose1 | 0 | 0
  Any Swelling, Prevenar13, Dose1 | 33 | 21
  Grade3 Swelling, Prevenar13, Dose1 | 1 | 0
  Any Erythema, GSK1437173A, Dose2: number analyzed (Participants) | 444 | 458
  Any Erythema, GSK1437173A, Dose2 | 147 | 128
  Grade3 Erythema, GSK1437173A, Dose2: number analyzed (Participants) | 444 | 458
  Grade3 Erythema, GSK1437173A, Dose2 | 9 | 5
  Any Pain, GSK1437173A, Dose2: number analyzed (Participants) | 444 | 458
  Any Pain, GSK1437173A, Dose2 | 326 | 359
  Grade3 Pain, GSK1437173A, Dose2: number analyzed (Participants) | 444 | 458
  Grade3 Pain, GSK1437173A, Dose2 | 28 | 32
  Any Swelling, GSK1437173A, Dose2: number analyzed (Participants) | 444 | 458
  Any Swelling, GSK1437173A, Dose2 | 70 | 72
  Grade3 Swelling, GSK1437173A, Dose2: number analyzed (Participants) | 444 | 458
  Grade3 Swelling, GSK1437173A, Dose2 | 1 | 2
  Any Erythema, GSK1437173A, Dose3: number analyzed (Participants) | 0 | 459
  Any Erythema, GSK1437173A, Dose3 | 0 | 123
  Grade3 Erythema, GSK1437173A, Dose3: number analyzed (Participants) | 0 | 459
  Grade3 Erythema, GSK1437173A, Dose3 | 0 | 1
  Any Pain, GSK1437173A, Dose3: number analyzed (Participants) | 0 | 459
  Any Pain, GSK1437173A, Dose3 | 0 | 350
  Grade3 Pain, GSK1437173A, Dose3: number analyzed (Participants) | 0 | 459
  Grade3 Pain, GSK1437173A, Dose3 | 0 | 41
  Any Swelling, GSK1437173A, Dose3: number analyzed (Participants) | 0 | 459
  Any Swelling, GSK1437173A, Dose3 | 0 | 60
  Grade3 Swelling, GSK1437173A, Dose3: number analyzed (Participants) | 0 | 459
  Grade3 Swelling, GSK1437173A, Dose3 | 0 | 0

7. Secondary Outcome: Number of Days With Each Solicited Local Symptoms
Description: The number of days with any local symptoms had been assessed during the post-vaccination period.
Time Frame: Within 7 days (Day 1 - 7) after each vaccination
Population: Analysis was performed on ES which included all subjects with at least one vaccine administration documented and who provided solicited safety data and for those who experienced the specified symptom for the specific dose.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 347 | 359
Days
  Any erythema,Dose1: number analyzed (Participants) | 131 | 31
  Any erythema,Dose1 | 3 [2 to 5] | 2 [1 to 4]
  Any pain,Dose1: number analyzed (Participants) | 347 | 241
  Any pain,Dose1 | 3 [2 to 4] | 2 [1 to 2]
  Any swelling, Dose1: number analyzed (Participants) | 76 | 21
  Any swelling, Dose1 | 2 [2 to 4] | 2 [1 to 3]
  Any erythema, Dose2: number analyzed (Participants) | 147 | 128
  Any erythema, Dose2 | 3 [2 to 4] | 2 [2 to 4]
  Any pain,Dose2: number analyzed (Participants) | 326 | 359
  Any pain,Dose2 | 3 [2 to 4] | 3 [2 to 4]
  Any swelling, Dose2: number analyzed (Participants) | 70 | 72
  Any swelling, Dose2 | 3 [2 to 4] | 2 [1.5 to 4]
  Any erythema,Dose3: number analyzed (Participants) | 0 | 123
  Any erythema,Dose3 |  | 2 [2 to 3]
  Any pain,Dose3: number analyzed (Participants) | 0 | 350
  Any pain,Dose3 |  | 3 [2 to 3]
  Any swelling,Dose3: number analyzed (Participants) | 0 | 60
  Any swelling,Dose3 |  | 2 [1 to 4]

8. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as oral temperature ≥ 38.0 degrees Celsius (°C)/ 100.4 degrees Fahrenheit (°F)], GastroIntestinal (GI) symptoms, headache, myalgia and shivering. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within 7 days (Day 1 - 7) after each vaccination
Population: Analysis was performed on ES which included all subjects with at least one vaccine administration documented and who provided solicited safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 448 | 463
Participants
  Any Fatigue, Dose1 | 166 | 85
  Grade3 Fatigue, Dose1 | 21 | 5
  Related Fatigue, Dose1 | 149 | 67
  Any Fever, Dose1 | 10 | 2
  Grade3 Fever, Dose1 | 1 | 0
  Related Fever, Dose1 | 8 | 0
  Any GI symptoms, Dose1 | 61 | 37
  Grade3 GI symptoms, Dose1 | 6 | 1
  Related GI symptoms, Dose1 | 55 | 30
  Any Headache, Dose1 | 130 | 72
  Grade3 Headache, Dose1 | 10 | 0
  Related Headache, Dose1 | 113 | 59
  Any Myalgia, Dose1 | 168 | 102
  Grade3 Myalgia, Dose1 | 17 | 4
  Related Myalgia, Dose1 | 150 | 86
  Any Shivering, Dose1 | 78 | 7
  Grade3 Shivering, Dose1 | 9 | 0
  Related Shivering, Dose1 | 71 | 7
  Any Fatigue, Dose2: number analyzed (Participants) | 444 | 458
  Any Fatigue, Dose2 | 192 | 152
  Grade3 Fatigue, Dose2: number analyzed (Participants) | 444 | 458
  Grade3 Fatigue, Dose2 | 22 | 17
  Related Fatigue, Dose2: number analyzed (Participants) | 444 | 458
  Related Fatigue, Dose2 | 177 | 141
  Any Fever, Dose2: number analyzed (Participants) | 444 | 458
  Any Fever, Dose2 | 16 | 7
  Grade3 Fever, Dose2: number analyzed (Participants) | 444 | 458
  Grade3 Fever, Dose2 | 2 | 2
  Related Fever, Dose2: number analyzed (Participants) | 444 | 458
  Related Fever, Dose2 | 10 | 2
  Any GI symptoms, Dose2: number analyzed (Participants) | 444 | 458
  Any GI symptoms, Dose2 | 57 | 47
  Grade3 GI symptoms, Dose2: number analyzed (Participants) | 444 | 458
  Grade3 GI symptoms, Dose2 | 8 | 4
  Related GI symptoms, Dose2: number analyzed (Participants) | 444 | 458
  Related GI symptoms, Dose2 | 50 | 44
  Any Headache, Dose2: number analyzed (Participants) | 444 | 458
  Any Headache, Dose2 | 156 | 115
  Grade3 Headache, Dose2: number analyzed (Participants) | 444 | 458
  Grade3 Headache, Dose2 | 18 | 7
  Related Headache, Dose2: number analyzed (Participants) | 444 | 458
  Related Headache, Dose2 | 143 | 99
  Any Myalgia, Dose2: number analyzed (Participants) | 444 | 458
  Any Myalgia, Dose2 | 203 | 174
  Grade3 Myalgia, Dose2: number analyzed (Participants) | 444 | 458
  Grade3 Myalgia, Dose2 | 23 | 24
  Related Myalgia, Dose2: number analyzed (Participants) | 444 | 458
  Related Myalgia, Dose2 | 186 | 163
  Any Shivering, Dose2: number analyzed (Participants) | 444 | 458
  Any Shivering, Dose2 | 95 | 50
  Grade3 Shivering, Dose2: number analyzed (Participants) | 444 | 458
  Grade3 Shivering, Dose2 | 12 | 8
  Related Shivering, Dose2: number analyzed (Participants) | 444 | 458
  Related Shivering, Dose2 | 86 | 47
  Any Fatigue, Dose3: number analyzed (Participants) | 0 | 459
  Any Fatigue, Dose3 | 0 | 210
  Grade3 Fatigue, Dose3: number analyzed (Participants) | 0 | 459
  Grade3 Fatigue, Dose3 | 0 | 27
  Related Fatigue, Dose3: number analyzed (Participants) | 0 | 459
  Related Fatigue, Dose3 | 0 | 202
  Any Fever, Dose3: number analyzed (Participants) | 0 | 459
  Any Fever, Dose3 | 0 | 23
  Grade3 Fever, Dose3: number analyzed (Participants) | 0 | 459
  Grade3 Fever, Dose3 | 0 | 2
  Related Fever, Dose3: number analyzed (Participants) | 0 | 459
  Related Fever, Dose3 | 0 | 17
  Any GI symptoms, Dose3: number analyzed (Participants) | 0 | 459
  Any GI symptoms, Dose3 | 0 | 69
  Grade3 GI symptoms, Dose3: number analyzed (Participants) | 0 | 459
  Grade3 GI symptoms, Dose3 | 0 | 3
  Related GI symptoms, Dose3: number analyzed (Participants) | 0 | 459
  Related GI symptoms, Dose3 | 0 | 63
  Any Headache, Dose3: number analyzed (Participants) | 0 | 459
  Any Headache, Dose3 | 0 | 180
  Grade3 Headache, Dose3: number analyzed (Participants) | 0 | 459
  Grade3 Headache, Dose3 | 0 | 23
  Related Headache, Dose3: number analyzed (Participants) | 0 | 459
  Related Headache, Dose3 | 0 | 168
  Any Myalgia, Dose3: number analyzed (Participants) | 0 | 459
  Any Myalgia, Dose3 | 0 | 224
  Grade3 Myalgia, Dose3: number analyzed (Participants) | 0 | 459
  Grade3 Myalgia, Dose3 | 0 | 37
  Related Myalgia, Dose3: number analyzed (Participants) | 0 | 459
  Related Myalgia, Dose3 | 0 | 215
  Any Shivering, Dose3: number analyzed (Participants) | 0 | 459
  Any Shivering, Dose3 | 0 | 122
  Grade3 Shivering, Dose3: number analyzed (Participants) | 0 | 459
  Grade3 Shivering, Dose3 | 0 | 20
  Related Shivering, Dose3: number analyzed (Participants) | 0 | 459
  Related Shivering, Dose3 | 0 | 117

9. Secondary Outcome: Number of Days With Solicited General Symptoms
Description: The number of days with any general symptoms had been assessed during the post-vaccination period. Assessed solicited general symptoms were fatigue, fever, GastroIntestinal (GI) symptoms, headache, myalgia and shivering.
Time Frame: Within 7 days (Day 1 - 7) after each vaccination
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 203 | 224
Days
  Any fatigue,Dose1: number analyzed (Participants) | 166 | 85
  Any fatigue,Dose1 | 2 [1 to 3] | 2 [1 to 3]
  Any GI symptoms,Dose1: number analyzed (Participants) | 61 | 37
  Any GI symptoms,Dose1 | 2 [1 to 2] | 1 [1 to 2]
  Any headache,Dose1: number analyzed (Participants) | 130 | 72
  Any headache,Dose1 | 2 [1 to 3] | 1 [1 to 2]
  Any myalgia,Dose1: number analyzed (Participants) | 168 | 102
  Any myalgia,Dose1 | 2 [1 to 3] | 2 [1 to 3]
  Any shivering,Dose1: number analyzed (Participants) | 78 | 7
  Any shivering,Dose1 | 1 [1 to 2] | 1 [1 to 3]
  Any fever,Dose1: number analyzed (Participants) | 10 | 2
  Any fever,Dose1 | 1 [1 to 1] | 1 [1 to 1]
  Any fatigue,Dose2: number analyzed (Participants) | 192 | 152
  Any fatigue,Dose2 | 2 [1 to 3] | 2 [1 to 3]
  Any GI symptoms,Dose2: number analyzed (Participants) | 57 | 47
  Any GI symptoms,Dose2 | 1 [1 to 2] | 1 [1 to 2]
  Any headache,Dose2: number analyzed (Participants) | 156 | 115
  Any headache,Dose2 | 2 [1 to 3] | 2 [1 to 3]
  Any myalgia,Dose2: number analyzed (Participants) | 203 | 174
  Any myalgia,Dose2 | 2 [1 to 3] | 2 [1 to 3]
  Any shivering,Dose2: number analyzed (Participants) | 95 | 50
  Any shivering,Dose2 | 1 [1 to 2] | 1 [1 to 2]
  Any fever,Dose2: number analyzed (Participants) | 16 | 7
  Any fever,Dose2 | 1 [1 to 1] | 1 [1 to 3]
  Any fatigue,Dose3: number analyzed (Participants) | 0 | 210
  Any fatigue,Dose3 |  | 2 [1 to 3]
  Any GI symptoms,Dose3: number analyzed (Participants) | 0 | 69
  Any GI symptoms,Dose3 |  | 1 [1 to 2]
  Any headache,Dose3: number analyzed (Participants) | 0 | 180
  Any headache,Dose3 |  | 1.5 [1 to 2]
  Any myalgia,Dose3: number analyzed (Participants) | 0 | 224
  Any myalgia,Dose3 |  | 2 [1 to 3]
  Any shivering,Dose3: number analyzed (Participants) | 0 | 122
  Any shivering,Dose3 |  | 1 [1 to 2]
  Any fever,Dose3: number analyzed (Participants) | 0 | 23
  Any fever,Dose3 |  | 1 [1 to 1]

10. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AE)
Description: An unsolicited AE covered any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 30 days (Day 1 to 30) after each vaccination
Population: Analysis was performed on ES which included all subjects with at least one vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 449 | 463
Participants
  Subjects with any AEs | 95 | 107
  Subjects with Grade 3 AEs | 9 | 13
  Subjects with related AEs | 35 | 25

11. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAE) From Day 1 to 30 Days Post Last Vaccination
Description: SAEs assessed included medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity. Related SAEs= SAEs assessed by the investigator as causally related to the study vaccination.
Time Frame: From first vaccination at Day 1 up to 30 days post last vaccination
Population: Analysis was performed on ES which included all subjects with at least one vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 449 | 463
Participants
  Subjects with any SAEs | 7 | 8
  Subjects with related SAEs | 0 | 0

12. Secondary Outcome: Number of Subjects With Any and Related SAEs From 30 Days Post Last Vaccination up to Study End.
Description: Serious adverse events (SAEs) assessed included medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity. Related SAEs= SAEs assessed by the investigator as causally related to the study vaccination.
Time Frame: From 30 days post last vaccination up to study end (Month 14 for the Co-Ad group and Month 16 for the Control group)
Population: Analysis was performed on ES which included all subjects with at least one vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 449 | 463
Participants
  Subjects with any SAEs | 10 | 10
  Subjects with related SAEs | 0 | 0

13. Secondary Outcome: Number of Subjects With Any and Related Potential Immune-mediated Diseases (pIMDs) From Day 1 to 30 Days Post Last Vaccination
Description: pIMDs assessed were a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which might or might not had an autoimmune aetiology. Related pIMDs= pIMDs assessed by the investigator as causally related to the study vaccination.
Time Frame: From first vaccination at Day 1 up to 30 days post last vaccination.
Population: Analysis was performed on ES which included all subjects with at least one vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 449 | 463
Participants
  Subjects with any pIMDs | 1 | 1
  Subjects with related pIMDs | 0 | 0

14. Secondary Outcome: Number of Subjects With Any pIMDs From 30 Days Post Last Vaccination up to Study End.
Description: pIMDs assessed were a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which might or might not had an autoimmune aetiology.
Time Frame: From 30 days post last vaccination up to study end (Month 14 for the Co-Ad group and Month 16 for the Control group)
Population: Analysis was performed on ES which included all subjects with at least one vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 449 | 463
Participants | 1 | 0

15. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms by Dose
Description: as for outcome 6
Time Frame: Within 7 days (Day 1 - 7) after each vaccination
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 448 | 463
Participants
  Any Erythema, Dose1 | 131 | 31
  Grade3 Erythema, Dose1 | 7 | 1
  Any Pain, Dose1 | 347 | 241
  Grade3 Pain, Dose1 | 28 | 9
  Any Swelling, Dose1 | 76 | 21
  Grade3 Swelling, Dose1 | 1 | 0
  Any Erythema, Dose2: number analyzed (Participants) | 444 | 458
  Any Erythema, Dose2 | 147 | 128
  Grade3 Erythema, Dose2: number analyzed (Participants) | 444 | 458
  Grade3 Erythema, Dose2 | 9 | 5
  Any Pain, Dose2: number analyzed (Participants) | 444 | 458
  Any Pain, Dose2 | 326 | 359
  Grade3 Pain, Dose2: number analyzed (Participants) | 444 | 458
  Grade3 Pain, Dose2 | 28 | 32
  Any Swelling, Dose2: number analyzed (Participants) | 444 | 458
  Any Swelling, Dose2 | 70 | 72
  Grade3 Swelling, Dose2: number analyzed (Participants) | 444 | 458
  Grade3 Swelling, Dose2 | 1 | 2
  Any Erythema, Dose3: number analyzed (Participants) | 0 | 459
  Any Erythema, Dose3 | 0 | 123
  Grade3 Erythema, Dose3: number analyzed (Participants) | 0 | 459
  Grade3 Erythema, Dose3 | 0 | 1
  Any Pain, Dose3: number analyzed (Participants) | 0 | 459
  Any Pain, Dose3 | 0 | 350
  Grade3 Pain, Dose3: number analyzed (Participants) | 0 | 459
  Grade3 Pain, Dose3 | 0 | 41
  Any Swelling, Dose3: number analyzed (Participants) | 0 | 459
  Any Swelling, Dose3 | 0 | 60
  Grade3 Swelling, Dose3: number analyzed (Participants) | 0 | 459
  Grade3 Swelling, Dose3 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs: During the 7-day (Days 1 to 7) after each vaccination, Unsolicited AEs: During the 30 day (Days 1 to 30) after any vaccination, SAEs: Throughout the study period [ Day 1 to study end (Month 14 for Co-Ad group and Month-16 for Control Group)]
Arm/Group | Co-Ad Group | Control Group
All-Cause Mortality (participants affected / at risk) | 2/449 | 4/463
Serious Adverse Events (participants affected / at risk) | 16/449 | 16/463
Other Adverse Events (participants affected / at risk) | 419/449 | 427/463
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Ad Group (N=449) | Control Group (N=463)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (2)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Ad Group (N=449) | Control Group (N=463)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pseudolymphoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Presbyacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 102 (118) | 119 (153)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue eruption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Administration site pruritus (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 139 (174) | 143 (179)
Fatigue (General disorders) | 243 (361) | 261 (448)
Feeling hot (General disorders) | 2 (2) | 2 (2)
Influenza like illness (General disorders) | 2 (2) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 192 (278) | 190 (286)
Injection site hypoaesthesia (General disorders) | 0 (0) | 1 (1)
Injection site movement impairment (General disorders) | 0 (0) | 1 (1)
Injection site oedema (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 389 (673) | 406 (952)
Injection site pruritus (General disorders) | 7 (9) | 7 (10)
Injection site rash (General disorders) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 1 (1)
Injection site swelling (General disorders) | 108 (146) | 117 (156)
Injection site warmth (General disorders) | 1 (1) | 2 (2)
Malaise (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 23 (26) | 29 (32)
Sensation of foreign body (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 5 (5) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 3 (3)
Injection site cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 7 (7)
Oral herpes (Infections and infestations) | 1 (1) | 2 (2)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 7 (7)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Mallet finger (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (10)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 260 (373) | 284 (501)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (3)
Headache (Nervous system disorders) | 206 (287) | 241 (376)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuromuscular blockade (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
VIth nerve paresis (Nervous system disorders) | 0 (0) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 6 (7) | 4 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Peau d'orange (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 5 (5)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT03439657/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT03439657/SAP_001.pdf